CLINICAL TRIAL: NCT01475773
Title: Impact of Personality Characteristics and Self-esteem on the Relationship Between Orthodontic Treatment Need and Oral-health Related Quality of Life in Adults.
Brief Title: Psychological Assessment of Adults Seeking Orthodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: ML7702
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-10

CONDITIONS: Self-esteem; Personality; Quality of Life; Malocclusion; Orthodontics
Keywords: self-esteem; personality; quality of life; malocclusion; orthodontics
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults (starting from age 17): adults seeking orthodontic treatment at the university of Leuven

SUMMARY:
Is their a association between the objective and subjective severity of a malocclusion, quality of life and self-esteem/personality (as modifier between objective/subjective severity and quality of life (cfr study Agou et al., 2008) ? A second goal is to compare motivation and expectations and the objective and subjective severity of the malocclusion on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* good health,
* thorough knowledge of the Dutch language

Exclusion Criteria:

* language

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: adults (starting from age 17) seeking orthodontic treatment on the first consultation of our clinic (university hospital Leuven)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Leuven, Leuven, Belgium

REFERENCES:
- [Background] Agou S, Locker D, Streiner DL, Tompson B. Impact of self-esteem on the oral-health-related quality of life of children with malocclusion. Am J Orthod Dentofacial Orthop. 2008 Oct;134(4):484-9. doi: 10.1016/j.ajodo.2006.11.021. PMID 18929265